CLINICAL TRIAL: NCT00225277
Title: A Double-Blind, Randomized, Comparator-Controlled Study In Subjects With Type 2 Diabetes Mellitus Comparing the Effects of Pioglitazone HCl Versus Glimepiride on the Rate of Progression of Coronary Atherosclerotic Disease as Measured by Intravascular Ultrasound
Brief Title: Efficacy Study of Pioglitazone Compared to Glimepiride on Coronary Atherosclerotic Disease Progression in Subjects With Type 2 Diabetes Mellitus
Acronym: PERISCOPE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 01-01-TL-OPI-516; U1111-1114-0400 (Registry Identifier: WHO)
Record Dates: First submitted 2005-09-21; First posted 2005-09-23 (Estimated); Results first posted 2009-06-10 (Estimated); Last update posted 2012-02-28 (Estimated); Status verified 2012-02

CONDITIONS: Diabetes Mellitus
Keywords: Glucose Metabolism Disorder; Dysmetabolic Syndrome; Type II Diabetes; Diabetes Mellitus, Lipoatrophic; Dyslipidemia; Drug Therapy; Atherosclerosis
MeSH Terms: conditions — Diabetes Mellitus; Glucose Metabolism Disorders; Diabetes Mellitus, Type 2; Diabetes Mellitus, Lipoatrophic; Dyslipidemias; Atherosclerosis | interventions — Pioglitazone; glimepiride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pioglitazone QD (Experimental)
  Interventions: Drug: Pioglitazone
- Glimepiride QD (Active Comparator)
  Interventions: Drug: Glimepiride

INTERVENTIONS:
Drug: Pioglitazone — Up to 45 mg pioglitazone (optimized for glucose control), tablets, orally, once daily for up to 72 weeks.
  Other Names: ACTOS®; AD4833
  Arms: Pioglitazone QD
Drug: Glimepiride — Up to 4 mg of glimepiride (optimized for glucose control), tablets, orally, once daily for up to 72 weeks.
  Arms: Glimepiride QD

SUMMARY:
The purpose of this study was to determine the efficacy of pioglitazone, once daily (QD), compared to glimepiride on atherosclerotic disease measured by intravascular ultrasound.

DETAILED DESCRIPTION:
Diabetes is a chronic disease with multiple metabolic defects that result in hyperglycemia arising from inadequate insulin activity. Type 2 diabetes is usually the result of a progression from reduced sensitivity of hepatic and peripheral tissue cells to circulating insulin (ie, insulin resistance) to a progressive inability of the body to produce adequate insulin to overcome insulin resistance (ie, insulin deficiency due to beta-cell insufficiency) resulting in impaired glucose tolerance and ultimately overt diabetes. In the United States, an estimated 21 million people have diabetes, with type 2 diabetes occurring in approximately 90% to 95% of cases. The goal of treating type 2 diabetes is to control blood glucose and thereby prevent long-term complications. Adequate glycemic control is paramount in attempting to avert chronic complications, including blindness; renal dysfunction resulting in dialysis or renal transplantation; neuropathy; non-traumatic amputations; and macrovascular complications, including myocardial ischemia and myocardial infarction, stroke, and peripheral arterial disease. Intensive glucose management in the early stages of diabetes may help forestall such complications.

Therapeutic agents have been developed to address each of the major functional metabolic defects associated with type 2 diabetes: decreased beta-cell function, elevated hepatic glucose output, and insulin resistance. Thiazolidinediones increase glucose utilization, decrease gluconeogenesis, and increase glucose disposal by binding to nuclear receptors known as peroxisome proliferator-activated receptors. Thiazolidinediones reduce insulin resistance by enhancing insulin sensitivity in muscle cells, adipose tissue, and hepatic cells (inhibiting hepatic gluconeogenesis), with no direct impact on insulin secretion. Thus, thiazolidinediones improve glycemic control and result in reduced levels of circulating insulin without predisposing patients to hypoglycemia. Peroxisome proliferator-activated receptors are found in tissues important for insulin action, such as adipose tissue, skeletal muscle, and the liver. The greatest concentration of peroxisome proliferator-activated receptors-gamma receptors is in adipose tissue.

This study was designed to compare the effects of pioglitazone compared to glimepiride on progression of atherosclerotic disease, as measured by intravascular ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* Females of childbearing potential who were sexually active agreed to use adequate contraception, and can neither be pregnant nor lactating from Screening throughout the duration of the study.
* Had a diagnosis of type 2 diabetes mellitus
* Have received appropriate counseling on lifestyle modification for type 2 diabetes, including diet and exercise.
* naïve to or was not currently taking antidiabetic therapy, or were currently treated with monotherapy or combination therapy.
* Had a glycosylated hemoglobin level greater than or equal to 6.0% and less than 9% at screening if taking antidiabetic medication or greater than or equal to 6.5% and less than 10% at screening if naive to or not taking antidiabetic medication.
* Angiographic criteria:

  * Entire Coronary Circulation: must have angiographic evidence of coronary heart disease as defined by at least 1 lesion in a native coronary artery that has greater than or equal to 20% reduction in lumen diameter by angiographic visual estimation.
  * Left Main Coronary Artery: must not have greater than 50% reduction in lumen diameter by visual angiographic estimation.
  * Target Coronary Artery:

    * The target vessel, which includes the main artery and all of its side branches, had not undergone prior percutaneous coronary intervention or coronary artery bypass graft surgery.
    * The target vessel, which includes the main artery and all of its side branches, was not currently a candidate for intervention or a likely candidate for intervention over the next 72 weeks.
    * The target vessel was not a bypass graft.
    * The target vessel was not infarct related.
* Had previous coronary artery bypass surgery at least six weeks prior to the qualifying intravascular ultrasound are eligible provided they are stable and meet all other entry criteria.
* Had an intravascular ultrasound tape deemed to be of acceptable intravascular ultrasound image quality and demonstrated adherence to the intravascular ultrasound interrogation protocol, as determined by the intravascular ultrasound Core Laboratory™ assessment.

Exclusion Criteria:

* Had type I diabetes mellitus.
* Had participated in another investigational study, or participated in an investigational study 30 days prior to the start of this study, or who were scheduled to participate in an investigational study during the time frame of this study.
* Male subjects who had a serum creatinine level greater than or equal to 2.0 mg/dL (greater than or equal to 177 µmol/L) (greater than or equal to 1.5 mg/dL; [greater than or equal to 133 µmol /L] if taking metformin) and female subjects who have serum creatinine greater than or equal to 1.8 mg/dL [greater than or equal to 159 µmol /L] (greater than or equal to 1.4 mg/dL [greater than or equal to 124 µmol /L] if taking metformin).
* Had unexplained microscopic hematuria greater than +1, confirmed by repeat testing.
* Had a history of drug abuse or a history of alcohol abuse (defined as regular or daily consumption of more than 4 alcoholic drinks per day) within the past 2 years.
* Had clinical cardiac failure as defined by New York Heart Association class III or IV, or known left ventricular dysfunction measured as left ventricular ejection fraction less than 40%, or by current use of diuretics or angiotensin converting enzyme inhibitors for treatment of heart failure.
* Had an alanine transaminase level of greater than 2.5 times the upper limit of normal active liver disease, or jaundice.
* Had a body mass index greater than 48 kg/m2 as calculated by weight (kg)/height (m2) or weight (pounds)/height (inches) 2 x 703.
* Was required to take or intended to continue taking any disallowed medication, any prescription medication, herbal treatment or over-the counter medication that may have interfered with evaluation of the study medication, including:

  * Chronically used oral glucocorticoids (eg, prednisone, cortisone, hydrocortisone, dexamethasone)
  * Niacin greater than100 mg a day, including niacin-containing products such as Advicor®
  * Chronically used steroid-joint injections
  * Thiazolidinediones
  * Sulfonylureas
  * Metformin/sulfonylurea combination
  * Other oral antidiabetic medications (eg, nateglinide [Starlix®], acarbose [Precose®]) with the exception of metformin
* Had known or suspected malignancy or recurrence of malignancy within the past 5 years, with the exception of basal cell carcinoma and Stage 1 squamous cell carcinoma of the skin.
* Had any disease where, in the opinion of the investigator (or designee), survival is expected to be less than 72 weeks.
* Clinical status was unstable (ie, requiring vasopressors or intravenous inotropes, intra-aortic balloon pump, hypotension [systolic blood pressure less than 90 mm Hg]).
* Prior to the screening visit, was scheduled for a staged cardiac intervention (percutaneous coronary intervention), peripheral vascular intervention, or coronary artery bypass graft surgery following the screening angiography.
* In the opinion of the investigator (or designee) had clinically significant valvular heart disease likely to require surgical repair/replacement during the course of the study.
* Had persistent, uncontrolled hypertension (ie, sitting systolic blood pressure greater than 160 mm Hg or sitting diastolic blood pressure greater than 100 mm Hg) at randomization.
* Males who had hemoglobin less than 10.5 g/dL (less than 105 g/L) and female subjects who had hemoglobin less than 10.0 g/dL (less than 100 g/L).
* Had a triglyceride level greater than 500 mg/dL (greater than 5.6 mmol/L).

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 547 (Actual)
Dates: Start 2003-07; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: VP Clinical Science, Study Director — Takeda
Locations (79):
- United States (65):
  - Birmingham, Alabama
  - Phoenix, Arizona
  - Huntington Beach, California
  - Los Angeles, California
  - Sacramento, California
  - San Diego, California
  - Torrance, California
  - Bridgeport, Connecticut
  - Farmington, Connecticut
  - Washington D.C., District of Columbia
  - Bay Pines, Florida
  - Jacksonville, Florida
  - Decatur, Georgia
  - Boise, Idaho
  - Chicago, Illinois
  - Edgewood, Kentucky
  - Lexington, Kentucky
  - Louisville, Kentucky
  - New Orleans, Louisiana
  - Bangor, Maine
  - Baltimore, Maryland
  - Detroit, Michigan
  - Flint, Michigan
  - Kalamazoo, Michigan
  - Petoskey, Michigan
  - Pontiac, Michigan
  - Royal Oak, Michigan
  - Ypsilanti, Michigan
  - Duluth, Minnesota
  - Minneapolis, Minnesota
  - Saint Cloud, Minnesota
  - Columbia, Missouri
  - Camden, New Jersey
  - Albany, New York
  - Mineola, New York
  - New York, New York
  - Rochester, New York
  - The Bronx, New York
  - Troy, New York
  - West Islip, New York
  - Williamsville, New York
  - Winston-Salem, North Carolina
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Columbus, Ohio
  - Westlake, Ohio
  - Oklahoma City, Oklahoma
  - Tulsa, Oklahoma
  - Abington, Pennsylvania
  - Bryn Mawr, Pennsylvania
  - Hershey, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Providence, Rhode Island
  - Greenville, South Carolina
  - Memphis, Tennessee
  - Oak Ridge, Tennessee
  - Amarillo, Texas
  - Houston, Texas
  - Lubbock, Texas
  - San Antonio, Texas
  - Charlottesville, Virginia
  - Norfolk, Virginia
  - Richmond, Virginia
  - Everett, Washington
  - Green Bay, Wisconsin
- Argentina (3):
  - Ciudad de Buenos Aires
  - Córdoba
  - Quilmes
- Canada (10):
  - Edmonton, Alberta
  - Vancouver, British Columbia
  - Victoria, British Columbia
  - Winnepeg, Manitoba
  - Saint John, New Brunswick
  - London, Ontario
  - Ottawa, Ontario
  - Montreal, Quebec
  - Sainte-Foy, Quebec
  - Saskatoon, Saskatchewan
- Santiago, Chile

REFERENCES:
- [Result] Nissen SE, Nicholls SJ, Wolski K, Nesto R, Kupfer S, Perez A, Jure H, De Larochelliere R, Staniloae CS, Mavromatis K, Saw J, Hu B, Lincoff AM, Tuzcu EM; PERISCOPE Investigators. Comparison of pioglitazone vs glimepiride on progression of coronary atherosclerosis in patients with type 2 diabetes: the PERISCOPE randomized controlled trial. JAMA. 2008 Apr 2;299(13):1561-73. doi: 10.1001/jama.299.13.1561. Epub 2008 Mar 31. PMID 18378631
- [Result] Betteridge DJ. CHICAGO, PERISCOPE and PROactive: CV risk modification in diabetes with pioglitazone. Fundam Clin Pharmacol. 2009 Dec;23(6):675-9. doi: 10.1111/j.1472-8206.2009.00741.x. Epub 2009 Sep 10. PMID 19744248
- [Result] Nicholls SJ, Tuzcu EM, Wolski K, Bayturan O, Lavoie A, Uno K, Kupfer S, Perez A, Nesto R, Nissen SE. Lowering the triglyceride/high-density lipoprotein cholesterol ratio is associated with the beneficial impact of pioglitazone on progression of coronary atherosclerosis in diabetic patients: insights from the PERISCOPE (Pioglitazone Effect on Regression of Intravascular Sonographic Coronary Obstruction Prospective Evaluation) study. J Am Coll Cardiol. 2011 Jan 11;57(2):153-9. doi: 10.1016/j.jacc.2010.06.055. PMID 21211686
- See also: ACTOS® Package Insert — http://general.takedapharm.com/content/file/pi.pdf?applicationcode=ab2d7112-8eb3-465a-8fda-35018a9eafb0&fileTypeCode=ACTOSPI

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled at 97 sites in the United States, Canada, Argentina and Chile from 21 July 2003 to 18 October 2007.
Pre-assignment Details: The participant flow results below do not include 4 subjects who were randomized but did not receive drug. Subjects participating in this study were enrolled in Pioglitazone or Glimepiride once daily (QD) treatment group.
Groups:
- Pioglitazone QD: Subjects received up to 45 mg Pioglitazone (dose optimized for glucose control) for up to 72 weeks.
- Glimepiride QD: Subjects received up to 4 mg Glimepiride (dose optimized for glucose control) for up to 72 weeks.
Period: Overall Study
Arm/Group | Pioglitazone QD | Glimepiride QD
Started | 274 (274 subjects randomized, but four subjects did not receive drug.) | 273 (Mean treatment durations were 56.3 weeks (glimepiride) and 56.5 weeks (pioglitazone).)
Completed | 177 | 178
Not Completed | 97 | 95
Not completed — Adverse Event | 30 | 34
Not completed — Lack of Efficacy | 4 | 1
Not completed — Lost to Follow-up | 4 | 6
Not completed — Physician Decision | 6 | 8
Not completed — Protocol Violation | 6 | 3
Not completed — Withdrawal by Subject | 40 | 34
Not completed — Other | 7 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pioglitazone QD | Glimepiride QD | Total
Number analyzed (Participants) | 270 | 273 | 543
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 189 | 193 | 382
  >=65 years | 81 | 80 | 161
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 84 | 93 | 177
  Male | 186 | 180 | 366
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 63 | 71 | 134
  Not Hispanic or Latino | 207 | 202 | 409
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Native American | 3 | 10 | 13
  Asian | 12 | 16 | 28
  Black or African American | 30 | 27 | 57
  White | 225 | 220 | 445
Family History of Coronary Artery Disease [Number; unit: Participants] — Was first degree male or female relative diagnosed with Coronary Artery Disease at age < 55 years or < 65 years, respectively?
  Participants
    Male Relative History | 91 | 77 | 168
    Female Relative History | 60 | 59 | 119
    No Family History | 119 | 137 | 256
Body Mass Index [Mean (Full Range); unit: Kg/m squared] — The mean for total was calculated as the weighted average of the means of the two treatment arms.
  Kg/m squared | 32.08 (5.264) [21.1 to 49.3] | 32.03 (5.233) [19.7 to 47.9] | 32.05 (0) [19.7 to 49.3]
Duration of Coronary Artery Disease [Mean (Full Range); unit: Months] — The mean for total was calculated as the weighted average of the means of the two treatment arms.
  Months | 40.4 (65.10) [0 to 378] | 40.5 (67.20) [0 to 468] | 40.4 (0) [0 to 468]
Duration of Diabetes Mellitus [Mean (Full Range); unit: Months] — The mean for total was calculated as the weighted average of the means of the two treatment arms.
  Months | 98.0 (100.25) [0 to 624] | 96.3 (89.51) [0 to 556] | 97.1 (0) [0 to 624]

OUTCOME MEASURES:

1. Primary Outcome: Nominal Change From Baseline in Percent Atheroma Volume
Description: The nominal change from baseline in percent atheroma volume for all slices of anatomically comparable segments of the target coronary artery. Assessment completed at the Week 72 visit or Final Visit if treatment was prematurely discontinued.
Time Frame: Baseline and Final Visit (up to 72 weeks)
Population: N at baseline included subjects who had both a baseline value and a final visit value. Baseline value is the last observation before first dose of study medication.
Measure: Least Squares Mean (Standard Error); unit: Percent volume
Arm/Group | Pioglitazone QD | Glimepiride QD
Number analyzed (Participants) | 179 | 181
Percent volume
  Baseline | 40.592 (0.6925) | 40.016 (0.6663)
  Nominal Change from Baseline | -0.161 (0.2095) | 0.725 (0.2017)
Statistical Analysis 1: Comparison: Pioglitazone QD vs Glimepiride QD; 2 Way analysis of covariance (ANCOVA), treatment and center effects with baseline value as covariate. Least Squares (LS) mean change and LS mean of the treatment difference reported; Test type: Superiority or Other; p = 0.002, ANCOVA; Mean Difference (Final Values) = -0.886, 95% CI [-1.4480 to -0.3250] — Mean Difference = Pioglitazone - Glimepiride

2. Secondary Outcome: Nominal Change From Baseline in Normalized Total Atheroma Volume
Description: The nominal change in normalized total atheroma volume as measured by the average of plaque areas for all slices of anatomically comparable segments of the target coronary artery multiplied by the mean number of matched slices in the population. Assessment completed at the Week 72 visit or Final Visit if treatment was prematurely discontinued.
Time Frame: Baseline and Final Visit (up to 72 weeks)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percent volume
Arm/Group | Pioglitazone QD | Glimepiride QD
Number analyzed (Participants) | 179 | 181
Percent volume
  Baseline | 206.579 (7.2778) | 217.619 (7.0030)
  Nominal Change from Baseline | -5.528 (1.5989) | -1.480 (1.5370)
Statistical Analysis 1: Comparison: Pioglitazone QD vs Glimepiride QD; 2 Way ANCOVA, treatment and center effects with baseline value as covariate. LS mean of the treatment difference reported; Test type: Superiority or Other; p = 0.064, ANCOVA; Mean Difference (Final Values) = -4.048, 95% CI [-8.3336 to 0.2374] — Mean Difference = Pioglitazone - Glimepiride

3. Secondary Outcome: Number of Subjects Experiencing Any of the Composite Endpoint A Cardiovascular Events
Description: Due to low event rates, number of subjects experiencing any of the composite endpoint A cardiovascular events is being reported instead of time to first occurrence. Endpoint A conditions listed in Limitations and Caveats section.
Time Frame: Up to 72 weeks
Population: Kaplan-Meier methodology was used to estimate time to event for each composite endpoint. P-value comparing survival function between groups was based on log-rank test. Time to first occurrence of cardiovascular events/hospitalizations had non-estimable medians due to very low event rates. Number of participants experiencing events are presented.
Measure: Number; unit: Participants
Arm/Group | Pioglitazone QD | Glimepiride QD
Number analyzed (Participants) | 270 | 273
Participants | 5 [0 to 0] | 6 [0 to 0]
Statistical Analysis 1: Comparison: Pioglitazone QD vs Glimepiride QD; Test type: Superiority or Other; p = 0.744, Log Rank — Kaplan-Meier methodology was used to estimate the time to event for each composite endpoint. The p-value was based on a log-rank test

4. Secondary Outcome: Number of Subjects Experiencing Any of the Composite Endpoint B Cardiovascular Events
Description: Due to low event rates, number of subjects experiencing any of the composite endpoint B cardiovascular events is being reported instead of time to first occurrence. Endpoint B conditions listed in Limitations and Caveats section.
Time Frame: Up to 72 weeks
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Pioglitazone QD | Glimepiride QD
Number analyzed (Participants) | 270 | 273
Participants | 40 [0 to 0] | 41 [0 to 0]
Statistical Analysis 1: Comparison: Pioglitazone QD vs Glimepiride QD; Test type: Superiority or Other; p = 0.883, Log Rank — [p-value comment as in outcome 3, analysis 1]

5. Secondary Outcome: Number of Subjects Experiencing Any of the Composite Endpoint C Cardiovascular Events
Description: Due to low event rates, number of subjects experiencing any of the composite endpoint C cardiovascular events is being reported instead of time to first occurrence. Endpoint C conditions listed in Limitations and Caveats section.
Time Frame: Up to 72 weeks
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Pioglitazone QD | Glimepiride QD
Number analyzed (Participants) | 270 | 273
participants | 11 [0 to 0] | 13 [0 to 0]
Statistical Analysis 1: Comparison: Pioglitazone QD vs Glimepiride QD; Test type: Superiority or Other; p = 0.663, Log Rank — [p-value comment as in outcome 3, analysis 1]

6. Other Pre Specified Outcome: Number of Cardiovascular Events as Adjudicated by the Clinical Endpoint Committee
Description: The incidence of cardiovascular events and composite endpoints occurring within 30 days of last dose as adjudicated by the Clinical Endpoint Committee. Abbreviations: PCI: Percutaneous Coronary Intervention; CABG: Coronary Artery Bypass Graft; CHF: Congestive Heart Failure.
Time Frame: Up to 72 weeks
Population: Safety Population
Measure: Number; unit: Number of Events
Arm/Group | Pioglitazone QD | Glimepiride QD
Number analyzed (Participants) | 270 | 273
Number of Events
  Nonfatal Myocardial Infarction | 2 | 4
  Nonfatal Stroke | 0 | 1
  Coronary Revascularization: PCI/CABG counted once | 29 | 30
  Coronary Revascularization: PCI | 25 | 28
  Coronary Revascularization: CABG | 5 | 2
  Carotid Endarterectomy/Stenting | 1 | 0
  Hospitalization for Unstable Angina | 4 | 2
  CHF Hospitalization: new/exacerbated counted once | 4 | 5
  Hospitalization for New CHF | 4 | 2
  Hospitalization for Exacerbated CHF | 0 | 3
  Noncardiovascular Mortality | 0 | 1
  Cardiovascular Mortality | 3 | 1
  Composite Endpoint A | 5 | 6
  Composite Endpoint B | 40 | 41
  Composite Endpoint C | 11 | 13

ADVERSE EVENTS:
Arm/Group | Pioglitazone QD | Glimepiride QD
Serious Adverse Events (participants affected / at risk) | 76 | 77
Other Adverse Events (participants affected / at risk) | 226 | 225
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Pioglitazone QD | Glimepiride QD
Abdominal Hernia (Gastrointestinal disorders) | 0/270 | 1/273
Abdominal Pain (Gastrointestinal disorders) | 1/270 | 1/273
Abdominal Strangulated Hernia (Gastrointestinal disorders) | 1/270 | 0/273
Accident at Work (Injury, poisoning and procedural complications) | 1/270 | 0/273
Acute Coronary Syndrome (Cardiac disorders) | 0/270 | 3/273
Acute Myocardial Infarction (Cardiac disorders) | 2/270 | 1/273
Acute Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 1/270 | 0/273
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/270 | 1/273
Anaemia (Blood and lymphatic system disorders) | 1/270 | 0/273
Anal Haemorrhage (Gastrointestinal disorders) | 0/270 | 1/273
Angina Pectoris (Cardiac disorders) | 8/270 | 4/273
Angina Unstable (Cardiac disorders) | 4/270 | 3/273
Aortic Stenosis (Vascular disorders) | 1/270 | 0/273
Appendiceal Mucocoele (Gastrointestinal disorders) | 0/270 | 1/273
Appendicitis Perforated (Gastrointestinal disorders) | 1/270 | 0/273
Astma (Respiratory, thoracic and mediastinal disorders) | 0/270 | 2/273
Atrial Fibrillation (Cardiac disorders) | 2/270 | 1/273
Atrioventricular Block Complete (Cardiac disorders) | 0/270 | 1/273
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 0/270 | 2/273
Biliary Colic (Hepatobiliary disorders) | 0/270 | 1/273
Bipolar II Disorder (Psychiatric disorders) | 0/270 | 1/273
Bladder Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/270 | 1/273
Blood Creatinine Increased (Investigations) | 0/270 | 1/273
Bronchitis (Infections and infestations) | 1/270 | 2/273
Bronchitis Acute (Infections and infestations) | 1/270 | 0/273
Cardiac Arrest (Cardiac disorders) | 0/270 | 1/273
Cardiac Discomfort (Cardiac disorders) | 0/270 | 1/273
Cardiac Failure Congestive (Cardiac disorders) | 3/270 | 5/273
Cardiac Tamponade (Cardiac disorders) | 0/270 | 1/273
Carotid Artery Stenosis (Nervous system disorders) | 1/270 | 0/273
Catheter Site Phlebitis (General disorders) | 1/270 | 0/273
Cellulitis (Infections and infestations) | 1/270 | 2/273
Cerebrospinal Fluid Leakage (Injury, poisoning and procedural complications) | 1/270 | 0/273
Cerebrovascular Accident (Nervous system disorders) | 0/270 | 1/273
Cerebrovascular Stenosis (Nervous system disorders) | 0/270 | 1/273
Cervical Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 1/270 | 0/273
Chloelithiasis (Hepatobiliary disorders) | 1/270 | 0/273
Cholecystitis (Hepatobiliary disorders) | 1/270 | 0/273
Cholecystitis Acute (Hepatobiliary disorders) | 0/270 | 1/273
Chronic Obstructive Airways Disease Exacerbated (Respiratory, thoracic and mediastinal disorders) | 0/270 | 3/273
Colitis (Gastrointestinal disorders) | 0/270 | 1/273
Constipation (Gastrointestinal disorders) | 0/270 | 1/273
Coronary Arterial Stent Insertion (Surgical and medical procedures) | 1/270 | 0/273
Coronary Artery Atherosclerosis (Cardiac disorders) | 1/270 | 1/273
Coronary Artery Disease (Cardiac disorders) | 20/270 | 16/273
Coronary Artery Insufficiency (Cardiac disorders) | 0/270 | 1/273
Coronary Artery Occlusion (Cardiac disorders) | 0/270 | 1/273
Coronary Artery Stenosis (Cardiac disorders) | 5/270 | 5/273
Costochondritis (Musculoskeletal and connective tissue disorders) | 0/270 | 1/273
Dehydration (Metabolism and nutrition disorders) | 1/270 | 0/273
Device Malfunction (Injury, poisoning and procedural complications) | 1/270 | 0/273
Diabetes Mellitus Inadequate Control (Metabolism and nutrition disorders) | 0/270 | 1/273
Diabetic Foot (Metabolism and nutrition disorders) | 1/270 | 0/273
Diabetic Foot Infection (Infections and infestations) | 0/270 | 1/273
Diverticulitis (Infections and infestations) | 1/270 | 2/273
Dizziness (Nervous system disorders) | 0/270 | 1/273
Dysphagia (Gastrointestinal disorders) | 1/270 | 0/273
Fall (Injury, poisoning and procedural complications) | 0/270 | 1/273
Flank Pain (Musculoskeletal and connective tissue disorders) | 1/270 | 0/273
Gastroenteritis (Infections and infestations) | 0/270 | 1/273
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0/270 | 1/273
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 1/270 | 0/273
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0/270 | 1/273
Hepatic Function Abnormal (Hepatobiliary disorders) | 0/270 | 1/273
Hepatitis (Hepatobiliary disorders) | 0/270 | 1/273
Hepatitis C Antibody Positive (Investigations) | 1/270 | 0/273
Hyperaldosteronism (Endocrine disorders) | 1/270 | 0/273
Hyperglycaemia (Metabolism and nutrition disorders) | 1/270 | 0/273
Hyperthyroidism (Endocrine disorders) | 1/270 | 0/273
Hypoclycaemia (Metabolism and nutrition disorders) | 0/270 | 3/273
Hypotension (Vascular disorders) | 1/270 | 0/273
Implant Site Infection (Infections and infestations) | 1/270 | 0/273
Incisional Hernia (Injury, poisoning and procedural complications) | 0/270 | 1/273
Intermittent Claudication (Vascular disorders) | 0/270 | 1/273
Interstitial Lung Disease (Respiratory, thoracic and mediastinal disorders) | 0/270 | 1/273
Ligament Injury (Injury, poisoning and procedural complications) | 0/270 | 1/273
Lobar Pneumonia (Infections and infestations) | 1/270 | 0/273
Localized Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1/270 | 1/273
Mental Disorder (Psychiatric disorders) | 1/270 | 0/273
Mental Status Changes (Psychiatric disorders) | 0/270 | 1/273
Myocardial Infarction (Cardiac disorders) | 3/270 | 2/273
Nasal Sinus Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/270 | 0/273
Non-Cardia Chest Pain (General disorders) | 15/270 | 5/273
Non-Small Cell Lung Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/270 | 0/273
Nystagmus (Nervous system disorders) | 1/270 | 0/273
Obesity (Metabolism and nutrition disorders) | 1/270 | 0/273
Oesophageal Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/270 | 1/273
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2/270 | 0/273
Peripheral Vascular Disorder (Vascular disorders) | 1/270 | 1/273
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1/270 | 0/273
Pneumonia (Infections and infestations) | 0/270 | 5/273
Pneumonia Primary Atypical (Infections and infestations) | 0/270 | 1/273
Post Procedural Haematoma (Injury, poisoning and procedural complications) | 1/270 | 0/273
Post Procedural Haemorrhage (Injury, poisoning and procedural complications) | 1/270 | 1/273
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 1/270 | 0/273
Renal Cell Carcinoma Stage Unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/270 | 0/273
Renal Failure (Renal and urinary disorders) | 0/270 | 1/273
Road Traffic Accident (Injury, poisoning and procedural complications) | 0/270 | 1/273
Ruptured Diverticulum of Colon (Gastrointestinal disorders) | 0/270 | 1/273
Small Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/270 | 1/273
Spinal Column Stenosis (Musculoskeletal and connective tissue disorders) | 1/270 | 0/273
Syncope (Nervous system disorders) | 1/270 | 1/273
Synovial Cyst (Metabolism and nutrition disorders) | 0/270 | 1/273
Therapeutic Agent Toxicity (Injury, poisoning and procedural complications) | 1/270 | 0/273
Upper Respiratory Tract Infection (Infections and infestations) | 0/270 | 1/273
Urinary Tract Infection (Infections and infestations) | 1/270 | 1/273
Ventricular Fibrillation (Cardiac disorders) | 1/270 | 0/273
Ventricular Tachycardia (Cardiac disorders) | 1/270 | 0/273
Vertigo (Ear and labyrinth disorders) | 1/270 | 0/273
Wound Infeciton (Infections and infestations) | 1/270 | 0/273
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Pioglitazone QD | Glimepiride QD
Angina Pectoris (Cardiac disorders) | 12/270 | 30/273
Arthralgia (Musculoskeletal and connective tissue disorders) | 17/270 | 15/273
Diarrhoea (Gastrointestinal disorders) | 11/270 | 14/273
Dizziness (Nervous system disorders) | 26/270 | 20/273
Fatigue (General disorders) | 17/270 | 14/273
Headache (Nervous system disorders) | 19/270 | 17/273
Hyperglycaemia (Metabolism and nutrition disorders) | 15/270 | 16/273
Hypertension (Vascular disorders) | 13/270 | 24/273
Hypoglycaemia (Metabolism and nutrition disorders) | 41/270 | 100/273
Influenza (Infections and infestations) | 14/270 | 9/273
Nasopharyngitis (Infections and infestations) | 13/270 | 22/273
Nausea (Gastrointestinal disorders) | 16/270 | 18/273
Non-Cardiac Chest Pain (General disorders) | 21/270 | 27/273
Oedema Peripheral (General disorders) | 48/270 | 30/273
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 15/270 | 19/273
Upper Respiratory Tract Infection (Infections and infestations) | 15/270 | 16/273
Urinary Tract Infection (Infections and infestations) | 17/270 | 19/273
Weight Increased (Investigations) | 28/270 | 15/273

LIMITATIONS AND CAVEATS:
Composite Endpoints A,B,C include cardiovascular mortality, nonfatal MI and nonfatal stroke. In addition, B: coronary revascularization, carotid endarterectomy/stenting, unstable angina hosp. or CHF; C: hospitalization for unstable angina or CHF.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review results communications prior to public release and can embargo trial results communications up to 150 days to permit actions necessary to preserve sponsor's intellectual property. Sponsor can request changes to the results communication only for the purpose of removing non study related information that is proprietary and confidential to sponsor. Sponsor can require delay of a results communication until the study has been completed at all participating sites.